CLINICAL TRIAL: NCT07066761
Title: Safety and Performance of a Pelvic Floor Mesh Implant for Laparoscopic Lateral Suspension (LatGYNious)
Brief Title: Safety and Performance of a Pelvic Floor Mesh Implant (LatGYNious)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.M.I. Agency for Medical Innovations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-52_001_LatGYNious; EUDAMED No: CIV-24-09-049116 (Other: EU (European Commission))
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse (POP); Genital Prolapse; Uterus Prolapse; Laparoscopic Surgery
Keywords: Laparoscopic lateral suspension (LLS)
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse | interventions — Surgical Mesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic lateral suspension with LatGYNious (with uterus preservation or after hysterectomy) (Active Comparator)
  Interventions: Device: Laparoscopic lateral suspension with surgical mesh (LatGYNious)

INTERVENTIONS:
Device: Laparoscopic lateral suspension with surgical mesh (LatGYNious) — Laparoscopic lateral suspension with LatGYNious (with uterus preservation or after hysterectomy)
  Other Names: surgical POP treatment; Pelvic organ prolapse

SUMMARY:
The purpose of the clinical investigation is to verify that the investigational device (LatGYNious) is appropriate to significantly improve the pelvic organ prolapse in patients.

DETAILED DESCRIPTION:
LatGYNious is a preformed mesh implant which combines two types of polypropylene meshes with different properties. The mesh body is made of ultra-light monofilament polypropylene with a wide hexagonal pore structure with a high level of elasticity. A reinforced mesh material with a smaller pore structure is used for the mesh arms, which achieves a strong lateral fixation. The overlap area of the two mesh types is designed to combine the properties of both structures. In case of a uterus preserving approach, the posterior part of the mesh body is removed.

The aim of the present study is to generate clinical data to show the safety and performance of LatGYNious for the treatment of female pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic prolapse in one of the 3 compartments from grade 2 with or without uterus
* Subject is candidate for a surgical treatment of pelvic organ prolapse
* Subject is willing and able to cooperate with follow-up examinations
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form and provided authorization to use and disclose information for research purposes.

Exclusion Criteria:

* Previous surgical treatment with a mesh implant for pelvic organ prolapse (mesh implant in anterior or posterior compartment)
* Active immunotherapy which may negatively affect the treatment with a surgical mesh
* Active cancer of the vagina / cervix / rectum
* . known or suspected hypersensitivity to Polypropylene
* Pregnancy
* participation in another study at the same time
* Unable to understand study requirements or is unable to comply with follow-up schedule
* Contraindicated according to the instruction for use of the device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Objective success | During follow-up until 6 and 12 months after surgery
  The primary objective is to confirm the effectiveness and objective success rate (anatomical correction defined by POP-Q) of a laparoscopic lateral mesh implant.
  Objective success is determined by anatomical measurement (POP-Q) pre- and post-operatively.
  Objective cure is defined as:
  * POP-Q values Ba, C and Bp < -1 (according to Barber et al.).
  * Absence of pelvic floor prolapse/bulge symptoms based on questionnaire (P-QoL).
  * No additional POP treatment necessary

SECONDARY OUTCOMES:
Quality of Life (QoL) | During follow-up until 6 and 12 months after surgery
  Quality of Life is determined by a validated questionnaire (P-QoL).
  The P-QoL Total score ranging from 0 points (complete continence) to 24 points (complete incontinence). An intra-individual comparison of preOP data vs. postOP data will be performed (for each follow-up).
Subjective success | During follow-up until 6 and 12 months after surgery
  Subjective rating of pelvic floor function is determined by a validated questionnaire (Deutscher Beckenboden-Fragebogen / German Pelvic Floor Questionnaire (GPFQ)).
  The GPFQ consist of 42 items, where each item has its scores. The scores were summed up for each category (bladder max. 45, bowel max. 34, prolapse max. 15, sexual max. 21).
  The final score were calculated as follows:
  (achieved value of category/ max. value of category)*10 Therefore, the max. value is 10 for each category and the final score is maximum 40.
  An intra-individual comparison of preOP data vs. postOP data will be performed (for each follow-up).
Complications | From operation during follow-up until 6 and 12 months after surgery.
  All adverse events will be reported.
  Serious device- and procedure-related adverse events will be summarized separately.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cadenbach-Blome, Dr. med., Principal Investigator — Medizincampus Bodensee - Klinik Tettnang
Locations (5):
- Austria (2):
  - BZK St. Johann in Tirol, Sankt Johann in Tirol, Tyrol
  - LKH Feldkirch, Gynäkologie und Geburtshilfe, Feldkirch
- Germany (3):
  - Universitätsklinik Brandenburg a.d. Havel, Klinik für Frauenheilkunde und Geburtshilfe, Brandenburg
  - Krankenhaus St. Joseph-Stift Bremen, Bremen
  - Medizincampus Bodensee - Klinik Tettnang, Tettnang

IPD SHARING:
Plan to Share IPD: No